CLINICAL TRIAL: NCT04692935
Title: Comparative Genomic Profiling of Lung Adenocarcinoma in Asians and Caucasians: A Propensity Matched Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jun Wang (Other)
Collaborators: Berry Genomics Co., Ltd. (Industry); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Jun Wang, Professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: 2020PHB375
Record Dates: First submitted 2020-12-25; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma of Lung
Keywords: Lung adenocarcinoma; Next-generation sequencing; Tumor genomic profiling; Ethnic differences
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asian lung adenocarcinoma: Asian LUADs patients who had broad-panel next-generation sequencing (NGS) performed on their primary tumor between January 2018 and December 2019 at the department of thoracic surgery of Peking University People's Hospital
- Caucasian lung adenocarcinoma: Caucasian LUADs patients who had targeted NGS (Memorial Sloan Kettering-Integrated Mutation Profiling of Actionable Cancer Targets [MSK-IMPACT]) will be identified in the AACR GENIE database, which consists of 6673 primary lung adenocarcinoma samples with clinical annotations

SUMMARY:
Lung adenocarcinomas (LUADs) from Asian ancestry are reported to have different genomic architectures compared with LUADs from Caucasian ancestry. However, due to lack of available cases, few studies controlled the clinical attributes during the comparisons of the genomic alterations. In this study, the investigators will identify Asian LUADs patients who had broad-panel next-generation sequencing (NGS) performed on their primary tumor between January 2018 and December 2019 at the department of thoracic surgery of Peking University People's Hospital. Then, Caucasian LUADs patients who had targeted NGS (Memorial Sloan Kettering-Integrated Mutation Profiling of Actionable Cancer Targets [MSK-IMPACT]) will be identified in the GENIE database, which consists of 6673 primary lung adenocarcinoma samples with clinical annotations. Finally, genomic alterations regarding somatic mutations, copy number variations, fusions, mutational signatures, oncogenic pathways, and therapeutic actionability will be comprehensively compared between these two cohorts after adjusting age, sex, smoking status, and pathologic stage using propensity score matching. This study will elucidate important ancestry differences between Asian and Caucasian lung adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung adenocarcinoma
* Broad-panel next-generation sequencing
* Asian

Exclusion Criteria:

* Inadequate clinicopathological information
* Low-quality next-generation sequencing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian LUADs patients who had broad-panel next-generation sequencing (NGS) performed on their primary tumor between January 2018 and December 2019 at the department of thoracic surgery of Peking University People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Oncoprint of somatic mutations | July 2021
  Association between genomic features and race
Copy number variations (CNVs) | July 2021
  CNVs analysis by race
Mutational signatures | August 2021
  Analysis of mutational signatures by race
Oncogenic pathways | September 2021
  Analysis of oncogenic pathways by race
Therapeutic actionability | October 2021
  Analysis of actionable alterations by race

IPD SHARING:
Plan to Share IPD: Undecided